CLINICAL TRIAL: NCT06519318
Title: Validity And Reliability of The Incremental Shuttle Walk Test In Individuals With Type 2 Diabetes Mellitus
Brief Title: Validity And Reliability of The Incremental Shuttle Walk Test In Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Ilayda Kayapinar (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Bezmialem Vakif University (Other)
Responsible Party: Sponsor-Investigator, Ilayda Kayapinar, Research Assistant, Istanbul Rumeli University
Organization: Istanbul Rumeli University (Other)
Other Study IDs: 2024/272
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus; Reliability and Validity
Keywords: Diabetes Mellitus; 6-Minute Walk Test; Incremental Shuttle Walk Test; Reliability and Validity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study was to determine the validity and reliability of the incremental shuttle walk test (ISWT) in patients with type 2 diabetes mellitus.This study involves the evaluation of the validity and test-retest reliability of the ISWT.

The assessments will be performed in two separate time periods. At the first visit, baseline assessments of the patient will be performed. These assessments include the recording of demographic information and the ISWT and 6 minute walk test assessments. Both tests will be performed with a 30-minute interval between them.

A retest will be performed 1 week after the initial assessment.

DETAILED DESCRIPTION:
Diabetes mellitus is a hormonal, metabolic and chronic disease characterised by hyperglycaemia resulting from a partial or complete deficiency of the hormone insulin or a defect in insulin-sensing receptors. Functional capacity is a vital marker for many chronic diseases, including Type 2 diabetes. Many things about the mechanism of decreased functional capacity specific to individuals with type 2 diabetes have not yet been clarified. As a result of the researches, it has been concluded that the deterioration in functional capacity is mostly related to glycaemic control and complications.

The Incremental Shuttle Walk Test (ISWT) is a maximal test that is widely used for the assessment of functional capacity and exercise tolerance because it is low cost and easy to perform. The incremental speed shuttle walk test was first described in 1992 to assess exercise capacity in patients with COPD. Compared to other field tests, ISWT is recommended because it shows high levels of maximum oxygen uptake (peak VO2) and provides physiological results closest to cardiopulmonary exercise testing (CPET), which is considered as the gold standard in the assessment of functional capacity.

The aim of our study was to determine the validity and reliability of the increasing speed shuttle walking test in patients with type 2 diabetes mellitus.

This study involves the evaluation of the validity and test-retest reliability of the ISWT.

The assessments will be performed in two separate time periods. At the first visit, baseline assessments of the patient will be performed. These assessments include the recording of demographic information and the ISWT and 6 minute walk test assessments. Both tests will be performed with a 30-minute interval between them.

A retest will be performed 1 week after the initial assessment.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c between 6.5 and 11
* No mental problems
* Able to walk independently

Exclusion Criteria:

* Lack of co-operation
* Uncontrolled diabetes,
* Patients with uncontrolled hypotension or hypertension
* Unstable cardiovascular and pulmonary conditions
* Having vertigo and various vestibular system disorders
* Those with severe neurological or severe respiratory diseases
* Patients with major musculoskeletal problems
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test | 15 minute
  For the reliability of the incremental shuttle walk test at the retest will be performed in 1 week. It is a field test consisting of 12 levels in which walking speed is increased. It is based on the principle of walking with an acceleration at an increasing speed in the up and down direction by passing around the cones on a 10-meter track with a distance of 9 metres between two cones by accepting turns around the cones as 0.5 meters. The distance covered is recorded during the test period. The increase in speed every minute is determined by three consecutive signals and only verbal warnings are given so that the individual can catch up with the speed during the test. If the individual is unable to continue the test (reaching maximal heart rate, pain, SpO2 value <80% extreme dyspnoea, fatigue), the test is terminated and the distance is recorded.

SECONDARY OUTCOMES:
Six Minute Walking Test | 10 minute
  The validity of the incremental shuttle test will be determined by 6 minute walking test. The test is performed in a thirty metre corridor. The distance walked over 30 meters for 6 minutes is recorded. Heart rate, dyspnoea level using the Borg scale, blood pressure and oxyhaemoglobin saturation can be determined before and after the test.

CONTACTS AND LOCATIONS:
Overall Officials: Melis USUL, RA, Principal Investigator — Istanbul Kent Universty; Gülenay YILDIRIM, RA, Principal Investigator — Istanbul Galata Universty; Gökşen KURAN ASLAN, Prof, Study Director — Istanbul Universty-Cerrahpaşa; Semiramis Özyılmaz, Assoc Prof, Study Director — Bezmaialem Foundation University; Muhammed TUNÇ, Asst Prof, Principal Investigator — Bezmaialem Foundation University
Locations (1):
- Bezmialem Foundation University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No